CLINICAL TRIAL: NCT06279247
Title: Proteomics and Metabolomics of Body Fluid in Patients With Narcolepsy
Status: Recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: KYLL-202212-011
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-11

CONDITIONS: Narcolepsy
Keywords: Narcolepsy; metabonomics; proteomics
MeSH Terms: conditions — Narcolepsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Information of subjects' medical records (basic information, scale score, sleep data, imaging examination) (10KB/ sample), collection of body fluid (blood (3ml/ case)/urine (3ml/ case)/stool (2g/ case)/cerebrospinal fluid (3ml/ case) from narcolepsy patients) Basic information (10KB/ sample), body fluids (blood (3ml/ case)/urine (3ml/ case)/stool (2g/ case)) of healthy subjects were collected (cerebrospinal fluid was not collected from healthy subjects).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- narcolepsy group
- health control group

SUMMARY:
Narcolepsy (NRL) is a rare chronic central nervous system dysfunction disease, which is more common in children and adolescents, and less common in adults. Its typical clinical features include excessive daytime sleep, paroxysmal cataplexy, sleep paralysis and sleep hallucination. In addition to the above typical manifestations, patients with narcolepsy can also manifest as hyperappetite, weight gain, multiple dreams, sleep fragmentation, anxiety and depression and other emotional disorders. In particular, in narcolepsy type 1 with cataplexy, cataplexy episodes can be confused with falls caused by seizures, transient ischemic attacks or neuromuscular disorders, or even mental conversion disorders. Due to its diverse clinical symptoms, it is easy to be missed and misdiagnosed.

At present, the pathogenesis of narcolepsy is still unclear, and its pathogenesis may be related to immune, genetic, environmental, infection, central nervous system degeneration and other factors. This study aims to investigate the changes of body fluid proteomics and metabolomics in patients with narcolepsy, and to provide an important basis for the pathogenesis of narcolepsy.

DETAILED DESCRIPTION:
1. Study design The baseline proteomics and metabolomics analysis of body fluid of narcolepsy (type 1 and type 2) and healthy volunteers, and the proteomics and metabolomics analysis of body fluid of narcolepsy patients after drug treatment were performed, and the differential metabolites and differential protein spots that could be used as potential molecular markers of narcolepsy were found by cross-sectional study.
2. Study subjects Source of study subjects: inpatients/healthy volunteers (Study subjects were well matched in gender, age, physical condition, etc.).
3. Study variables (factors) and measurements 3.1 Data collected from all subjects included: medical record information (basic information, scale score, sleep data, imaging examination) (10KB/ sample), body fluid (blood (3ml/ case)/urine (3ml/ case)/stool (2g/ case)/cerebrospinal fluid (3ml/ case) collected from narcolepsy patients).

Basic information (10KB/ sample), body fluids (blood (3ml/ case)/urine (3ml/ case)/stool (2g/ case)) of healthy subjects were collected (cerebrospinal fluid was not collected from healthy subjects).

Baseline proteomic and metabolomics assays were performed. Proteomics and metabolomics of body fluid in narcolepsy patients after drug treatment. (Sample collection requires metabolomics sampling in the same season and time period) 3.2 Assessment of sleepiness

1. Sleepiness assessment: Epworth sleepiness scale (ESS), Pittsburgh sleep quality index (PSQI)
2. Diagnostic evaluation of sleepiness: sleep apnea monitoring (PSG) and multiple sleep latency test (MSLT) were completed. Overnight polysomnography (PSG) can provide detailed physiological sleep information and multiple sleep latency test (MSLT) can objectively measure sleepiness. The multiple Sleep latency testing experiment (MSLT) was performed the day after an overnight PSG recording that showed ≥ 6 hours of adequate sleep at night and could effectively explain the MSLT data. The MSLT was based on 20-min PSG recordings that were repeated every 2 h, 4-5 times per day, starting approximately 2 h after morning awakening. Individuals were asked to attempt to fall asleep at each time point. The ICSD-3 states that in order to diagnose narcolepsy, the mean sleep latency of MSLT should be 8 minutes or less and more than two sleep-onset rapid eye movement periods (SOREMPs).

Study outcomes

1. omics analysis of metabolic mechanisms related to narcolepsy and screening of co-enriched pathways. To screen potential molecular markers related to the biological characteristics and prognosis of narcolepsy.
2. To study the body fluid and imaging characteristics of narcolepsy patients. 5. Data collection and management Data collection was performed using a paper case report form, and subject information (basic information, scale scores, sleep data, imaging examination) was entered into a computer by someone. Baseline proteomics and metabolomics of body fluid (blood/urine/stool/cerebrospinal fluid) in patients with narcolepsy (type 1 and type 2) and body fluid (blood/urine/stool) in healthy volunteers. Proteomics and metabolomics of body fluid in narcolepsy patients after drug treatment. Statistical analysis was performed by a clinical statistician.

ELIGIBILITY:
Inclusion Criteria

* All patients met the diagnostic criteria of the International Classification of Sleep Disorders, Third edition (ICSD-3).

Exclusion Criteria

* primary hypersomnia or hypersomnia due to shift work, sleep deprivation and other sleep rhythm disturbances;
* excessive sleep due to drug abuse;
* suffering from Parkinson's disease, Alzheimer's disease and other nervous system diseases and mental diseases;
* complicated with heart, lung, liver, kidney, blood endocrine system and other basic diseases, or acute chronic infection in a short period of time;
* Use of sedatives, hypnotics, antidepressants, lithium and dopamine receptor antagonists for two weeks before examination;
* patients who cannot cooperate with PSG and MSLT due to various factors.

Ages: 5 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with narcolepsy
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-08-26 (Estimated); Study Completion 2025-08-26 (Estimated)

PRIMARY OUTCOMES:
To screen potential molecular markers related to the biological characteristics and prognosis of narcolepsy. | 2022.09~2024.09
  1. omics analysis of metabolic mechanisms related to narcolepsy and screening of co-enriched pathways. To screen potential molecular markers related to the biological characteristics and prognosis of narcolepsy.
  2. To study the body fluid and imaging characteristics of narcolepsy patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China